CLINICAL TRIAL: NCT05735119
Title: A Multi-Center, Prospective Post-Market Clinical Follow-Up Study: Subscapularis Repair Augmented With Tapestry Biointegrative Implant After Shoulder Arthroplasty Evaluation (RAISE)
Brief Title: Embody Post-Market Clinical Follow-Up Study
Acronym: RAISE
Status: Enrolling by invitation | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: EMBODY-003
Record Dates: First submitted 2023-02-06; First posted 2023-02-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Tendon Injuries- Subscapularis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subscapularis Tendon Injuries: Tapestry Biointegrative Implant
  Interventions: Device: Tapestry Biointegrative Implant

INTERVENTIONS:
Device: Tapestry Biointegrative Implant — Collagen-based implant composed of type I bovine collagen and poly(D,L-lactide). It is designed to function as a non-constricting, protective layer between the tendon and surrounding tissues. Preclinical studies of the Tapestry implant showed dense collagenous fibrous connective tissue ingrowth into and around the implant.

SUMMARY:
A multi-center, prospective post-market clinical follow-up study: subscapularis repair augmented with Tapestry Biointegrative Implant after shoulder arthroplasty. The primary objective of this study is to evaluate the long-term integrity of the subscapularis tendon repair after shoulder arthroplasty augmented with Tapestry Biointegrative Implant, assessed by ultrasound 6 months postoperatively. Secondary objectives are to assess shoulder function (internal rotation strength), safety, and patient reported outcomes. Patients will be evaluated preoperatively, at the time of surgery, 3, 6, 12 and 24 months after surgery.

DETAILED DESCRIPTION:
The proposed investigation is a multi-center, prospective patient registry: subscapularis repair augmented with TAPESTRY® Biointegrative Implant after shoulder arthroplasty. The primary objective of this study is to evaluate the long-term integrity of the subscapularis tendon repair after shoulder arthroplasty augmented with TAPESTRY Biointegrative Implant, assessed by ultrasound 6 months postoperatively. Secondary objectives are to assess shoulder function (internal rotation strength), safety, and patient reported outcomes. Patients will be evaluated preoperatively, at the time of surgery, 3, 6, 12 and 24 months after surgery. A total of 100 patients will be enrolled. Enrolled subjects will include adults undergoing shoulder arthroplasty, who meet the study eligibility criteria. The Tapestry Biointegrative Implant was FDA 510(k) cleared (K201572) on October 22, 2020, for the management and protection of tendon injuries in which there has been no substantial loss of tendon tissue. The primary analysis of subscapularis tendon repair integrity assessed by ultrasound will occur when all study subjects reach 6 months post-surgery. The goal of the analysis is to show that the tendon failure rate for subscapularis repair with Tapestry is lower than the failure rate for subscapularis repair without Tapestry a receiving surgery with the Tapestry and the literature-defined failure rate for tendon healing. Secondary endpoints will be analyzed when the last subject reaches the 24 month timepoint.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, 21 years and older.
2. Patient requires shoulder arthroplasty (anatomic or reverse) with subscapularis repair due to osteoarthritis, rotator cuff injury, rheumatoid arthritis and/or other inflammatory disorder, osteonecrosis, and/or post-traumatic injury (e.g., humerus fractures).
3. Patients healthy enough to undergo primary anatomic or reverse shoulder arthroplasty, in the opinion of the investigator;
4. Patients receiving shoulder arthroplasty with anticipated subscapularis tenotomy (ST) or subscapularis peel (SP).
5. Intact rotator cuff including subscapularis tendon for anatomic shoulder arthroplasty or a repairable subscapularis tendon for reverse shoulder arthroplasty, as determined by preoperative examination or imaging, if indicated or available preoperatively. Imaging is not required for this assessment.
6. Ability and willingness to comply with prescribed post-operative rehabilitation program.
7. Ability and willingness to comply with follow-up visit schedule.
8. Able to understand the informed consent process, including regulatory requirements such as HIPAA authorization, and document informed consent prior to completion of any study-related procedures.
9. Ability to read, understand, and complete subject-reported outcomes in English.

Exclusion Criteria:

1. Shoulder arthroplasty requiring a lesser tuberosity osteotomy or revision arthroplasty.
2. Prior index shoulder surgery requiring treatment to the subscapularis.
3. Intraoperative identification of irreparable subscapularis tear (rTSA)
4. Diabetic patients with hemoglobin A1c (HbA1c) level >8% prior to surgery.
5. Patients with inflammatory arthritis or patients that are immunocompromised, or patients that have a glenoid deficiency.
6. Patients with a known history of hypersensitivity to bovine-derived materials.
7. Hypersensitivity to poly(D,L-lactide) materials.
8. Females of child-bearing potential who are pregnant or plan to become pregnant during the course of the study.
9. Currently involved in any injury litigation or worker's compensation claims relating to the index shoulder.
10. Enrolled, or plans to enroll, in another clinical trial during this study that would affect the outcomes of this study.
11. History of non-compliance with medical treatment, physical therapy/rehabilitation, or clinical study participation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing shoulder arthroplasty, who meet the study eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Subscapularis repair integrity | 6 months postoperatively
  Assessed by ultrasound evaluation per the EMBODY-003 ultrasound procedure manual.

SECONDARY OUTCOMES:
Subscapularis tendon tissue quality | 6 months postoperatively
  Assessed using ultrasound to evaluate and measure thickness compared to normal (9, 10) subscapularis tendon thickness at 6-months postoperatively. Tendon tissue thickness and quality evaluation will be measured by trained personnel per the EMBODY-003 ultrasound procedure manual.
Internal rotation strength in the belly-press (11,12) position, measured by an electronic handheld dynamometer. | Screening visit/3 months postoperatively/6 months postoperatively/12 months postoperatively/24 months postoperatively
  Subscapularis repair integrity
Subscapularis repair integrity | Screening visit/3 months postoperatively/6 months postoperatively/12 months postoperatively/24 months postoperatively
  Assessed by internal rotation strength in the Bear-Hug position.
Adverse events | Surgery visit/3 months postoperatively/6 months postoperatively/12 months postoperatively/24 months postoperatively
  Procedure and/or treatment
Serious adverse events | Surgery visit/3 months postoperatively/6 months postoperatively/12 months postoperatively/24 months postoperatively
  Procedure and/or treatment
Serious adverse events necessitating a second surgical intervention (SSI) | Surgery visit/3 months postoperatively/6 months postoperatively/12 months postoperatively/24 months postoperatively
  Procedure and/or treatment
Patient Questionnaire | 3 months postoperatively/6 months postoperatively/12 months postoperatively/24 months postoperatively
  Patient Satisfaction
Forward evaluation | Screening visit/3 months postoperatively/6 months postoperatively/12 months postoperatively/24 months postoperatively
  Active Range of Motion (ROM)
Abduction | Screening visit/3 months postoperatively/6 months postoperatively/12 months postoperatively/24 months postoperatively
  Active ROM
External rotation | Screening visit/3 months postoperatively/6 months postoperatively/12 months postoperatively/24 months postoperatively
  Active ROM
Internal rotation | Screening visit/3 months postoperatively/6 months postoperatively/12 months postoperatively/24 months postoperatively
  Active ROM
American Shoulder and Elbow Surgeon Evaluation (ASES) | Baseline/3 months/6 months/12 months/24 months postoperatively
  Patient reported clinical outcome scores
Visual Analog Scale (VAS) | Screening visit/3 months postoperatively/6 months postoperatively/12 months postoperatively/24 months postoperatively
  Patient reported clinical outcome scores
Simple Shoulder Test (SST) | Screening visit/3 months postoperatively/6 months postoperatively/12 months postoperatively/24 months postoperatively
  Patient reported clinical outcome scores

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Alta Orthopaedics, Santa Barbara, California
  - HCA Florida - JFK Hospital, Atlantis, Florida
  - Atlantis Orthopaedics, Palm Beach Gardens, Florida
  - Central Indiana Orthopedics, Carmel, Indiana
  - University of Louisville Physicians, Inc., Louisville, Kentucky